CLINICAL TRIAL: NCT02715648
Title: Using Phenazopyridine for In-office Cystoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Urogynecology Associates (Other)
Responsible Party: Principal Investigator, Eman Elkadry, M.D., Principle Investigator, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 003-2016
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Cystoscopy; Phenazopyridine
MeSH Terms: interventions — Phenazopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Phenazopyridine before cystoscopy (No Intervention): This group will not receive phenazopyridine prior to cystoscopy
- Phenazopyridine before cystoscopy (Experimental): This group will receive 200mg of phenazopyridine prior to cystoscopy
  Interventions: Drug: Phenazopyridine

INTERVENTIONS:
Drug: Phenazopyridine
  Arms: Phenazopyridine before cystoscopy

SUMMARY:
The investigators propose to conduct a randomized controlled trial to evaluate whether administration of phenazopyridine prior to the procedure decreases office cystoscopy time. Women undergoing in-office cystoscopy at Boston Urogynecology will be recruited.

DETAILED DESCRIPTION:
All potentially eligible participants will have had a complete history, physical examination, urinalysis and urine culture for clinical purposes. After eligibility is confirmed and written, informed consent is obtained, participants will be randomized to one of the two study arms. Participants randomized to phenazopyridine arm will receive 200 mg by mouth approximately 60 minutes prior to the scheduled cystoscopy. During the cystoscopy, at various time points, the time will be recorded.The color of the efflux will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing in-office diagnostic cystoscopy at Boston Urogynecology Associates

Exclusion Criteria:

* Women who have taken vitamin B the day of the cystoscopy
* Cystoscopy with concurrent treatments such as botulinum toxin or periurethral bulking injections
* Allergy to phenazopyridine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Total cystoscopy time | at time of cystoscopy
  The total time of cystoscopy will be measured

SECONDARY OUTCOMES:
Time to visualization of ureteral jets | at time of cystoscopy
  The time to visualization of the first ureteral jet will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elkadry, MD, Principal Investigator — Practitioner
Locations (1):
- Boston Urogynecology Associates, 725 Concord Ave. Suite 1200, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No